CLINICAL TRIAL: NCT01183481
Title: Aprepitant and Granisetron for the Prophylaxis of Radiation Induced Nausea and Vomiting - A Pilot Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was stopped due to inadequate accrual.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Principal Investigator, Dr. Edward Chow, Professor, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RINV Prophylaxis
Record Dates: First submitted 2010-08-04; First posted 2010-08-17 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Nausea; Vomiting
Keywords: nausea; vomiting; antiemetics; radiotherapy; Radiation-induced nausea and vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Aprepitant; Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aprepitant and Granisetron (Experimental): Patients will be given a single dose of Granisetron 2 mg orally and Aprepitant 125 mg on Day 0 (at least one hour before on the day of RT) followed by 80 mg of Aprepitant once daily in the mornings on Days 1 and 2 following the Palliative radiation therapy.
  Interventions: Drug: Aprepitant; Radiation: Palliative radiation therapy; Drug: Granisetron

INTERVENTIONS:
Drug: Aprepitant — Patients will be given a single dose of Aprepitant 125 mg on Day 0 (at least one hour before on the day of RT) followed by 80 mg of Aprepitant once daily in the mornings on Days 1 and 2 following the radiation treatment.
Radiation: Palliative radiation therapy — Moderately emetogenic palliative radiation therapy (RT) will be administered to all patients on the study.
Drug: Granisetron — Patients will be given a single dose of both Granisetron 2 mg orally on Day 0 (at least one hour before on the day of RT).

SUMMARY:
The primary objective of this pilot study is to examine the efficacy of Aprepitant given in combination with Granisetron for the prevention of delayed-phase RINV in 84 patients receiving a single 8Gy of moderately emetogenic palliative RT in the RRRP at Sunnybrook Odette Cancer Centre for painful bony metastases from any primary solid tumor. Patients will be given a single dose of Granisetron 2 mg orally and Aprepitant 125 mg on Day 0 (at least one hour before on the day of RT) followed by 80 mg of Aprepitant once daily in the mornings on Days 1 and 2 following the radiation treatment.. Secondary objectives include determining the complete RINV prophylaxis rate (acute and delayed phases), the partial emesis control rate, the safety of the combined regime, QOL issues, the time to the first emetic event and the time to the first use of rescue medication .

ELIGIBILITY:
Inclusion Criteria:

* Patients with bone metastases from any primary solid tumor site scheduled to receive a single 8 Gy fraction of palliative radiotherapy considered to be moderately emetogenic (an area of at least 80 cm2 in the anterior/posterior direction and located between the level of upper border of T11 and the lower border of L3) in the RRRP at Sunnybrook Odette Cancer Centre will be considered eligible.

Exclusion Criteria:

* Exclusion criteria include having nausea or vomiting 24hrs prior to radiation
* Having received or being scheduled to receive cranial radiation, moderately or highly emetogenic cytotoxic therapy 7 days prior to, during, or after radiation, receiving corticosteroids (except inhaled or topical), 5HT3 receptor antagonists or NK-1 antagonists or other antiemetic medication, being allergic to study medications, having a KPS<40, being pregnant or of childbearing potential and not using contraceptive measures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Chow, MBBS PhD FRCPC, Principal Investigator — Odette Cancer Centre, Sunnybrook Health Sciences Centre
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between January 2011 and October 2012 in a radiation oncology clinic
Pre-assignment Details: No enrolled patients were later excluded.
Groups:
- Aprepitant and Granisetron: Patients will be given a single dose of Granisetron 2 mg orally and Aprepitant 125 mg on Day 0 (at least one hour before on the day of RT) followed by 80 mg of Aprepitant once daily in the mornings on Days 1 and 2 following the radiation treatment.
Period: Overall Study
Arm/Group | Aprepitant and Granisetron
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aprepitant and Granisetron
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (15.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 8
Region of Enrollment [Number; unit: participants]
  Canada | 19

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Experiencing no Vomiting and no Nausea, Without Use of Any Rescue Antiemetic Medication(s), From Days 2-10 Following the Radiation Therapy (Delayed RINV).
Description: Assessments of nausea, vomiting, and antiemetic use will be taken daily within 2-10 following the radiation therapy based on patient self-report nausea/vomiting diaries.
Time Frame: Days 2-10 following radiotherapy
Measure: Number; unit: participants
Arm/Group | Aprepitant and Granisetron
Number analyzed (Participants) | 19
participants | 19 [NA to NA]

2. Secondary Outcome: The Complete RINV Prophylaxis Rate (Acute and Delayed Phases), the Partial Emesis Control Rate, the Safety of the Combined Regime, QOL Issues, the Time to the First Emetic Event and Use of Rescue Medication .
Description: Data will be measured by research staff at baseline and patient self-report nausea diaries will be taken on each day within this time frame.
Time Frame: From day of radiotherapy to 10 days following radiotherapy
Reporting Status: Not Posted

3. Secondary Outcome: Control Rate of Acute Phase Nausea, Vomiting, and Retching in Patients Undergoing Single Fraction Radiotherapy
Description: Percentage of participants experiencing no nausea, vomiting, and retching during the acute phase was assessed.
  Assessments of nausea, vomiting, and antiemetic use will be taken daily following the radiation therapy based on patient self-report nausea/vomiting diaries.
Time Frame: Day of radiotherapy and 24 hours following
Population: Patients undergoing single fraction treatment
Measure: Number; unit: percentage of participants
Arm/Group | Aprepitant and Granisetron
Number analyzed (Participants) | 13
percentage of participants
  Control rate of acute phase nausea | 100
  Control rate of acute phase vomiting/retching | 100

4. Secondary Outcome: Control Rate of Delayed Phase Nausea, Vomiting, and Retching in Patients Undergoing Single Fraction Radiotherapy
Description: Percentage of participants in the single fraction arm experiencing no nausea, vomiting, and retching was assessed.
  Assessments of nausea, vomiting, and antiemetic use will be taken daily within 2-10 following the radiation therapy based on patient self-report nausea/vomiting diaries.
Time Frame: Days 2-10 following radiotherapy
Population: Patients undergoing single fraction treatment
Measure: Number; unit: percentage of participants
Arm/Group | Aprepitant and Granisetron
Number analyzed (Participants) | 13
percentage of participants
  Control rate of delayed phase nausea | 62
  Control rate of delayed phase vomiting/retching | 85

5. Secondary Outcome: Control Rate of Acute Phase Nausea, Vomiting, and Retching in Patients Undergoing Multiple Fraction Radiotherapy
Description: Percentage of participants in the multiple fraction arm experiencing no nausea, vomiting, and retching was assessed.
  Data will be measured by research staff at baseline and patient self-report nausea diaries will be taken on each day within this time frame.
Time Frame: During radiotherapy (5 days) and the 24 hours following radiotherapy
Population: Patients undergoing multiple fraction treatment
Measure: Number; unit: percentage of participants
Arm/Group | Aprepitant and Granisetron
Number analyzed (Participants) | 6
percentage of participants
  Control rate of acute phase nausea | 67
  Control rate of acute phase vomiting/retching | 67

6. Secondary Outcome: Control Rate of Delayed Phase Nausea, Vomiting, and Retching in Patients Undergoing Multiple Fraction Radiotherapy
Description: Percentage of participants experiencing no nausea, vomiting, and retching was assessed.
  Assessments of nausea, vomiting, and antiemetic use will be taken daily within 2-10 following the radiation therapy based on patient self-report nausea/vomiting diaries.
Time Frame: Days 2-10 following radiotherapy
Population: Patients undergoing multiple fraction treatment
Measure: Number; unit: percentage of participants
Arm/Group | Aprepitant and Granisetron
Number analyzed (Participants) | 6
percentage of participants
  Control rate of delayed phase nausea | 83
  Control rate of delayed phase vomiting/retching | 83

ADVERSE EVENTS:
Arm/Group | Aprepitant and Granisetron
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aprepitant and Granisetron (N=19)
Pain crisis (Musculoskeletal and connective tissue disorders) | 1 — One patient required admission to hospital for pain control following radiation planning, which was not attributable to the study intervention.

LIMITATIONS AND CAVEATS:
Small number of subjects results in early termination of study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No